CLINICAL TRIAL: NCT01122056
Title: Effect of Aerobic Exercise on Side Effects of Disease Modifying Therapy With Subcutaneous Interferon-b1b in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: H10-00277
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; b1b-interferon; Fatigue; Exercise
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A = Active group (Active Comparator): Patients will receive interactive exercise training session from an experienced multiple sclerosis
  Interventions: Other: Physical exercise training
- B = Control group (Placebo Comparator) (No Intervention): Patients will receive general advice about benefits/side effects of physical activity in multiple sclerosis.

INTERVENTIONS:
Other: Physical exercise training — Two 2-hours long interactive training to perform safe and efficient aerobic exercise for patients with multiple sclerosis
  Other Names: Betaseron b1b-interferon; Aerobic exercise
  Arms: A = Active group

SUMMARY:
The purpose of this study is to investigate the effects and tolerability of exercise on side effects of injectable disease modifying treatments in multiple sclerosis. The investigators main hypothesis is that controlled exercise is safe and can be well tolerated in patients with multiple sclerosis and it can improve disease modifying treatment related side effects such as fatigue.

DETAILED DESCRIPTION:
Patient compliance with disease modifying treatment largely depends on relatively common side effects of such treatments such as fatigue. Regular exercise can potentially improve these side effects. However, Safety and effects of exercise has not been studied in patients with multiple sclerosis. Our main aim is to study the safety, tolerability and effects of exercise on side effects of subcutaneous interferon-b1b in patients with Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of relapsing remitting multiple sclerosis on treatment with b1b-interferon disease modifying treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Multiple Sclerosis Fatigue
Quality of Life
Injection site visual analog scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Boyd, Study Director — University of British Columbia; Kristen Campbell, Study Director — University of British Columbia; Saul Isserow, Study Director — University of British Columbia
Locations (1):
- Vancouver Coastal Health: University of British Columbia Hospital, Vancouver, British Columbia, Canada